CLINICAL TRIAL: NCT07278986
Title: Single Dose Investigator Initiated Pilot Study to Investigate CYTALUX (Pafolacianine) for Intraoperative Imaging of Patients With Endometrial Cancer Planned for Surgery
Brief Title: CYTALUX for Intraoperative Imaging of Patients With Endometrial Cancer
Acronym: CYTALUX ISS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 22825
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer; Near Infrared Fluorescence Imaging; CYTALUX (Pafolacianine) Injection; Planned Diagnostic Laparoscopies
Keywords: Endometrial Cancer; Near Infrared Fluorescence Imaging; Cytalux (pafolacianine) injection; surgery; surgery planned; camera; investigational
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Intervention Model Description: This is a single center, single dose, open-label investigator-initiated pilot study in adult subjects with a primary diagnosis of endometrial cancer who are being evaluated for surgery. Subjects will receive one dose of CYTALUX™ (pafolacianine) injection intravenously prior to the planned diagnostic laparoscopies. This hour-long infusion will be completed from 1 hour to up to 168 hours (7 days) prior to intraoperative near-infrared (NIR) imaging for the planned surgery. All subjects participating in the study are expected to receive CYTALUX™ injection and standard care laparoscopic evaluation of disease. Intraoperative imaging with Cytalux will be performed for assessment of disease detection in patients who are being evaluated to undergo surgery for endometrial cancer. Any tissues removed as part of standard of care will undergo assessment with NIR light imaging prior to and after resection. This will be then compared to gold standard histologic confirmation by pathology.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CYTALUX™ (pafolacianine) injection and standard care laparoscopic evaluation of disease. (Other): single dose, open-label, pilot study of single dose of CYTALUX (pafolacianine) injection
  Interventions: Drug: CYTALUX™ (pafolacianine); Device: 1788 4K Camera System with Advanced Imaging Modality

INTERVENTIONS:
Drug: CYTALUX™ (pafolacianine) — CYTALUX™ (pafolacianine) injection and standard care laparoscopic evaluation of disease. Intraoperative imaging with Cytalux will be performed for assessment of disease detection in patients who are being evaluated to undergo surgery for endometrial cancer. Any tissues removed as part of standard of care will undergo assessment with NIR light imaging prior to and after resection. This will be then compared to gold standard histologic confirmation by pathology.
Device: 1788 4K Camera System with Advanced Imaging Modality — Combination Product

SUMMARY:
The research study is being done to assess the safety and ability of an investigational drug called CYTALUX (pafolacianine) and a special camera system for the detection of cancer in patients undergoing surgical resection for endometrial cancer.

DETAILED DESCRIPTION:
Study participant's medical history (questions about their health) will be reviewed with them before their surgery to ensure they are able to participate in the study.

It is important for study participants to tell their doctor if they are taking vitamins that contain Folic Acid (vitamin B9), or Folic Acid (vitamin B9) supplements. They will need to stop taking these vitamins at least 48 hours before their scheduled infusion. Folic acid can reduce the effectiveness of the CYTALUX (pafolacianine). Certain other medications have not been studied together with CYTALUX (pafolacianine), so it is important for them to tell their doctor about all medicines and supplements they are taking.

Screening Visit (To see if they can take part in the study and will take place no more than 30 days before surgery)

The following will take place during the Screening Visit. These tests could include those that their doctor would do before any major surgery, in which case they may not be repeated for this trial.

• The doctor and/or a member of the doctor's team will ask them about their health, and obtain a list of all medications, including vitamins and over-the-counter medications (medicines obtained without a doctor's prescription), that they are taking.

Study Drug Infusion (Up to 7 days before surgery)

* Study participants will be scheduled to receive the drug being tested, CYTALUX (pafolacianine), any time from 7 days before their surgery up to the day of their surgery. They will receive CYTALUX (pafolacianine) at least one hour before the imaging portion of their surgery.
* Before they receive the study drug, the following will happen:

  * The doctor and/or a member of the doctor's team will ask about their health and obtain a list of all medications including vitamins and over-the-counter (medicines obtained without a doctor's prescription) medicines that they are taking.
  * For patients who are able to have children, a urine pregnancy test will be done.
* The study drug will be given over about 60 minutes through a vein. The dose of CYTALUX (pafolacianine) given will be calculated by their weight.

Surgery Visit

The following activities related to the study will happen on the day of surgery:

* The doctor will look for cancer as they usually do by feeling and looking throughout the peritoneal cavity using white light and will record the findings.
* After this, the doctor will use the special camera system to look for cancer that may light up where the CYTALUX (pafolacianine) has attached and will record the findings. Any cancer that is seen with the use of the special camera system may be the same as what the doctor recorded earlier without the use of the camera system, or there may be additional cancer seen.
* The doctor will then remove the cancer that has been detected, and any areas that they think should be taken out. This removal of the cancer will be done as the doctor would usually do in surgery for endometrial cancer.
* After the doctor has removed the cancer as discussed above, she/he will once again use the camera system to see if there is any cancer left and the findings will be recorded. Any such cancer observed will be removed based on the doctor's judgment.
* The cancer tissue that is removed will be sent to the lab for further testing.
* Any side effects that a participant may have with the use of CYTALUX (pafolacianine) and/or the camera system will be recorded.
* A sample of any cancer that is removed during this study will be sent to the hospital's laboratory for testing to see if it is endometrial cancer, and to see if the cancer has certain receptors on the surface that would cause the drug, CYTALUX (pafolacianine), to attach to the cancer.

Post-operation Visit (Day 28 ± 7 Days)

* About 4 weeks after the surgery, study participants will be contacted via phone by the doctor and/or a member of the doctor's team, or asked to come to the clinic.
* They will be asked about how they are feeling and about all the medications, including vitamins and over-the-counter (medicines obtained without a doctor's prescription) medicines, that they are taking. The findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Adult subjects 18 years of age and older
3. Primary diagnosis of endometrial cancer
4. Scheduled to undergo surgery for endometrial cancer
5. Ability to understand the requirements of the study and agree to abide by the study restrictions and to return for the required assessments
6. Willingness to stop the use of folate or folic acid supplements at least 48 hours prior to infusion of study drug

Exclusion Criteria:

1. Pregnancy or positive pregnancy test
2. Any medical condition that in the opinion of the investigator could potentially jeopardize the safety of the subject
3. History of anaphylactic reactions to products containing indocyanine green
4. History of allergy to any of the components of CYTALUX
5. Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol or follow-up schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-18 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 2 months after surgery
  The primary efficacy endpoint is the sensitivity of CYTALUX with NIR imaging for detection of malignant lesions. Sensitivity is defined as the proportion of fluorescent light positive lesions that are histologically confirmed to be cancer relative to the total number of lesions confirmed to be cancer.
  Sensitivity = (True Positive)/(True Positive + False Negative)

SECONDARY OUTCOMES:
Secondary Endpoints | 2 months after surgery
  1. Incidence rates of all adverse events (AEs), adverse device effects (ADEs), and SAEs, from the time of CYTALUX administration through Visit 3
  2. Sensitivity for cancerous lesions for:
     1. FRα positive lesions
     2. FRβ positive lesions

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Abramson Cancer Center at Penn Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania Gynecologic Oncology Department, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data will be shared without IPD.

DOCUMENTS (2):
  • Study Protocol (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT07278986/Prot_000.pdf
  • Informed Consent Form (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT07278986/ICF_001.pdf